CLINICAL TRIAL: NCT02972762
Title: The Clinical Investigation of Anesthesia Depth's Influence in Total Intravenous Anesthesia on Postoperative Delirium of Elderly Patients
Brief Title: Anesthesia Depth's Influence on Postoperative Delirium
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: XiangyaH
Record Dates: First submitted 2016-11-16; First posted 2016-11-23 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2016-11

CONDITIONS: Femur Head Necrosis
Keywords: depth of anesthesia\postoperation delirium
MeSH Terms: conditions — Femur Head Necrosis | interventions — Propofol

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- L Group (Active Comparator): The participants in L Group will receive Lumbar plexus and sciatic nerve block with ropivacaine before anesthesia induction.The investigator use Diprivan TCI target-controlled infusion during anesthesia induction period, target effect-site concentration is set at 4.0g / kg. After reaching the target concentration, sufentanil 0.2g / kg is administrated, Laryngeal mask will be placed into participant's mouth at 2 min after sufentanil is given. Anesthesia will be maintained with remifentanil TCI target-controlled infusion and Diprivan BIS close-loop target controlled infusion,BIS ranges from 50 to 60.The values of BP,P,PetCO2 will be controled in proper site. each participant will be given postoperative analgesia pump to release postoperative pain.
  Interventions: Drug: Diprivan
- D Group (Active Comparator): The participant in L Group will receive Lumbar plexus and sciatic nerve block with ropivacaine before anesthesia induction.The investigator use Diprivan TCI target-controlled infusion during anesthesia induction period, target effect-site concentration is set at 4.0g / kg. After reaching the target concentration, sufentanil 0.2g / kg is administrated, Laryngeal mask will be placed into participant's mouth at 2 min after sufentanil is given. Anesthesia will be maintained with remifentanil TCI target-controlled infusion and Diprivan BIS close-loop target controlled infusion,BIS ranges from 35 to 45.The values of BP,P,PetCO2 will be controled in proper site. The investigator use postoperative analgesia pump to control postoperative pain for each participant.
  Interventions: Drug: Diprivan

INTERVENTIONS:
Drug: Diprivan — anesthesia will be maintained with remifentanil and Diprivan.we use Diprivan close-loop to control the anesthesia depth,and the anesthesia depth will be detected with BIS machine.the usage of remifentanil、ropivacaine、sufentanil and cisatracurium in both arms is no difference.

SUMMARY:
The investigators,according to the eligibility criteria,plane to choose 80 elderly anticipates who will undergo selective hip replacement surgery.This participants will be randomly divided into 2 groups:light anesthesia depth group(L Group) and deep anesthesia depth group (D Group).Before anesthesia induction,each participant will be given lumbar plexus and sciatic nerve block in order to control pain of interoperative and postoperative.During operation period,the L Group will be kept in light anesthesia depth(BIS:50-60),while the D group will be kept in deep anesthesia depth(BIS:35-45)--The BIS values in the range of 30-60 have been recommended in general anesthesia.After operation,a PCIA(patient controlled intravenous analgesia) analgesia pump will be given to each participant to control postoperative pain. The investigator will evaluate the mental state of participant with MMSE(mini-mental state examination) before surgery and review each participant with a CAM-CR for 3 days after surgery to assess the situation of postoperation delirium.intraoperative awareness,postoperative pain will also be investigated in postoperative days 1, 2, 3.

DETAILED DESCRIPTION:
The investigators,according to the eligibility criteria,plane to choose 80 elderly participants who will undergo selective hip replacement surgery.This participants will be randomly divided into 2 groups:light anesthesia depth group(BIS:50-60) and deep anesthesia depth group (BIS:35-45)--The BIS values in the range of 30-60 have been recommended in general anesthesia.Before anesthesia induction,each participant will be given lumbar plexus and sciatic nerve block in order to control pain of intraoperative and postoperative.The investigator use propofol 4ug\kg、and sufentanil 0.2ug\kg during anesthesia induction period,after that,a Laryngeal mask will be placed into patient's mouth.Anesthesia is maintained with remifentanil TCI(target-controlled infusion) target-controlled infusion(concentration:2ng/ml) and propofol BIS closed-loop target-controlled infusion.During the operation period ,the investigator keep the L Group's BIS range from 50 to 60.While the D Group's BIS range from 35 to 45.All participants receive postoperative analgesia.After operation,all participants will be send to PACU(post-anaesthesia care unit ) to wake up and send back to ward,And a PCIA(patient controlled intravenous analgesia) analgesia pump will be given to each participants to control postoperative pain.The investigators will use MMSE(mini-mental state examination) to evaluate the participant's mental state before surgery.For 3 days after operation,The investigator will review each participant with a CAM-CR to assess the situation of postoperation delirium.The investigator will see if there is intraoperative awareness by asking questions.Postoperative pain(with VAS) will also be investigated in postoperative days 1, 2, 3.

ELIGIBILITY:
Inclusion Criteria:

1. participant who is selected to undergo hip replacement surgery.
2. participant who is older than 60 years old.
3. participant whose ASA（The American Society of Anesthesiologists） is II-III.
4. participant whose BMI is 18-25.
5. participant who is able to understand and complete The Confusion Assessment Method(CAM-CR).
6. participant who is able to finish Visual Analogue Scale(VAS).
7. participant who is conscious and willing to take part in this research.
8. participant and his/her relatives are willing to take part in this research.

Exclusion Criteria:

1. participant who has serious liver or kidney disease.
2. participant who suffer from mental or neurologic disease,such as Alzheimer disease.
3. participant who has undergone cardiovascular surgery or neurosurgery.
4. participant who has have sedation or antidepression medicine for a long time.
5. participant who has something wrong with his/her vision or hearing.
6. participant who has blood coagulation dysfunction.
7. participant who is an illiteracy.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
postoperative delirium score(with The Confusion Assessment Method) | 3 days
  the The Confusion Assessment Method is widely used to access the postoperative delirium all around the world.the total score more than 22 means that the The participant has got delirium.
final data analysis | 10 days
  the investigators use SPSS software to analysis data.

SECONDARY OUTCOMES:
postoperative pain score(with visual analogue scale) | 3 days
intraoperative awareness | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: tao Zhong, doctor, Study Director — Xiangya hospital of CSU
Locations (1):
- Xiangya hospital of CSU, Changsha, Hunan, China